## Official Title:

A Cognitive Self-Management Intervention for Persons with Multiple Sclerosis: Adapting Web-based Technology

## Statistical Analysis Plan

Results will be entered into a computer database for analysis using IBM SPSS Statistics version 25. Data will be checked for accuracy by research staff. Reliability estimates (internal consistency) will be determined for each instrument, and alphas of >0.70 will be considered acceptable. Descriptive analyses will be performed to obtain a description of the sample on demographic and illness-related variables. Analysis of covariance (ANCOVA) will be used to measure the differences between groups while controlling for continuous variables that might affect the outcome (e.g., age, length of diagnosis). The significance level for this pilot study will be alpha <0.10. Feasibility measures will look for trends in the data focusing on recruitment and retention of participants over the 8-week intervention, problems and solutions encountered using the web-based video conferencing platform by the interventionist and/or the participants, wear ability of the ActiGraph wrist watches for seven days.